## Consent form Phase 1 & 2 Retrospective sample follow up







### **Covid Response study (COVRES)**

### **Participant Consent Form**

**NCT XXX** 

09/07/2020

### Consent form Phase 1 & 2 Retrospective sample follow up









### Participant Consent Form Phase 1 & 2

**Study Title:** A Northern Ireland population study of SARS-CoV-2 prevalence, predisposing factors and pathology

| Participant Identification no: | | |
|---|---|---|
| Chief Investigator: Prof Tony Bjourson | <b>Phone:</b> (028)71 675 661 | Email: aj.bjourson@ulster.ac.uk |

#### Please confirm, by marking the boxes provided, that you agree with the following statements:

| 1. | I have been given and have read and understood the information sheet dated 09/07/2020 |
|---|---|
| | version 6 for the above study and have asked and received answers to any questions raised. |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time |
| | without giving any reason and without my rights being affected in any way. |
| 3. | I agree to the collection, processing and use of my biological samples and personal data for |
| | this study on the terms outlined in the Participant Information sheet and I understand that |
| | genomic data and data will be generated from my biological samples. |
| 4. | I understand that my paper and electronic medical records (including Northern Ireland |
| | Electronic Care Record (NIECR) and other NHS electronic systems) will hold relevant |
| | information to this study and I consent for members of the research team to access this |
| | information if required for one year to follow the progression of my condition. |
| 5. | I understand that the researchers will hold all information and data collected during the |
| | study securely and in confidence and that all efforts will be made to ensure that I cannot |
| | be identified as a participant in the study (except as might be required by law) and I |
| | consent for the researchers to hold relevant personal data |
| 6. | I understand that my pseudonymised data generated as part of this study will be retained |
| | indefinitely for scientific research purposes, in accordance with EU data protection laws |
| 7. | I consent to inclusion of my pseudonymised data in the Northern Ireland Centre for |
| | Stratified Medicine database. |
| 8. | I consent that in the event of loss of capacity on my behalf, any samples and personal |
| | information collected prior to this event will remain in the study and consent to |
| | continued follow-up of my clinical notes |
| 9. | I agree and consent to provide blood sample (s) for the purposes of this study and |
| | confirm that I have been given details of the amount(s) and time points that they are to |
| | be taken and how it will be stored, used and the method of disposal. |

# Consent form Phase 1 & 2 Retrospective sample follow up







| | | NO |
|---|---|---|
| 19 | Would you like your GP to be informed you are taking part in this research study? | YES |
| | I am under no obligation to take part in any future studies. | |
| | studies of a similar nature. I understand that I am agreeing only to receive information and | |
| 18. | I agree and consent to being contacted at a later date and invited to take part in future | |
| 17. | I agree and consent to take part in the above study | |
| | which they will be stored for 10 years | |
| | c. I do not wish my blood or tissues to be used for any purpose other than this study for | С. |
| | isolation of my genetic material <b>OR</b> | |
| | OR b. I consent to their indefinite storage and use in any future study that does not involve the | b. |
| | a. I consent to their indefinite storage and use in any future study including genetic studies, | |
| | studies have been explained to me and (Please read carefully and only tick one box): | |
| 16. | The potential benefits of keeping my blood or other tissues for future research | |
| 15. | I understand that I will not receive any individual results or feedback | |
| 14. | I understand that I will not be paid to take part in this study | |
| | commercial (for-profit) companies. | |
| | understand that the research organisations accessing pseudonymised data could include | |
| | pseudonymised clinical and biological data from my previously donated samples and I | |
| 13. | I agree and consent that approved research organisations can have access to | |
| | for secure processing and analysis. | |
| 12. | to Ulster University approved research organisations within or outside the UK, and EEA, | |
| 12. | I agree and consent that my donated sample(s), DNA, and associated data could be sent | |
| | Participant Information Sheet. | |
| | the data for research via a managed data access committee (DAC) as described in the | |
| 11. | data on the European <b>GISAID</b> database (where, researchers will have controlled access to | |
| 11. | will be stored, used and the method of disposal. I consent to the research team sharing a copy of my de-identified health data and genomic | |
| | been given details of the amount and time points that samples are to be taken and how it | |
| 10. | I agree to provide a saliva sample for the purposes of this study and confirm that I have | |

Appendix 3

# Consent form Phase 1 & 2 Retrospective sample follow up

Version 6 09/07/2020





| 1 |
|----------------------|
| Ulster<br>University |

| Name of Participant (please print) | Signature | Date (dd/mmm/yy) |
|------------------------------------|-----------|------------------|
| Name of Researcher | Signature | Date (dd/mmm/yy) |